CLINICAL TRIAL: NCT06533553
Title: An Open-label Phase II Study to Assess the Pharmacodynamic (PD) Effects of Dexpramipexole in Participants With Eosinophilic Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A Study to Assess the Effects of Dexpramipexole in Participants With Eosinophilic COPD
Acronym: SUSPIRE-1
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Areteia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AR-DEX-23-05
Record Dates: First submitted 2024-07-30; First posted 2024-08-01 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- 150 mg dexpramipexole BID (Experimental): 150 mg dexpramipexole oral tablet taken twice a day
  Interventions: Drug: Dexpramipexole Dihydrochloride

INTERVENTIONS:
Drug: Dexpramipexole Dihydrochloride — Administration of dexpramipexole tablet

SUMMARY:
This is an open-label Phase II study assessing the PD of dexpramipexole 150 mg twice daily (BID) in participants with eosinophilic COPD. This study will help characterize the profile and duration of reductions of blood absolute eosinophil counts (AEC).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form prior to any study-specific procedures.
* Male or female ≥40 to ≤80 years of age at Screening Visit.
* Physician diagnosis of COPD for at least 2 years prior to the Screening Visit in accordance with the definition by the American Thoracic Society/European Respiratory Society
* Current or former smokers with a cigarette smoking history of ≥10 pack years at the Screening Visit calculated as (number of pack years = [number of cigarettes per day/20] multiplied by number of years smoked). Former smokers are defined as those who meet the pack-year history but have stopped smoking for at least 6 months prior to the Screening Visit.
* Spirometry: post-BD FEV1/FVC <0.70 and post-BD FEV1 >20% and ≤60% of predicted normal values at the Screening Visit.
* Documented history of exacerbation risk defined as exacerbation history of ≥1 moderate* or ≥1 severe** within 2 years prior to the Screening Visit.
* Background ICS-based therapy (ICS+ long-acting β2 agonist [LABA], or ICS + long-acting muscarinic antagonist [LAMA], or ICS + LAMA + LABA) for ≥12 weeks prior to enrollment with a stable dose of medication for ≥4 weeks prior to the Screening Visit.
* Evidence of an eosinophilic phenotype: Participants with blood eosinophils ≥0.30x109/L at the Screening Visit.
* Negative urine pregnancy test for women of childbearing potential (WOCBP) at the Screening and Baseline Visits.
* WOCBP (after menarche) must use e methods of birth control from the Screening Visit through the End of Study Visit..

Exclusion Criteria:

* A current diagnosis of asthma or any history of asthma diagnosis when ≥40 years of age.
* Significant pulmonary disease other than COPD (eg, α-1 antitrypsin deficiency, active tuberculosis, lung fibrosis, sarcoidosis, interstitial lung disease, pulmonary hypertension, lung cancer, clinically significant bronchiectasis, Churg-Strauss Syndrome) or another diagnosed pulmonary or systemic disease associated with elevated eosinophil counts.
* Pneumonia, upper or lower respiratory tract infection or acute exacerbation of COPD within 4 weeks prior to or during the Screening Phase.
* Treatment with a biologic investigational drug in the last 5 months prior to the Screening Visit. Treatment with non-biologic investigational drugs in the previous 30 days or five-half-lives prior to the Screening Visit, whichever is longer. Treatment with GSK3511294 (long-acting anti-interleukin-5) in the past 12 months.
* Treatment with any of the following monoclonal antibody therapies within 120 days prior to the Baseline Visit: benralizumab, dupilumab, mepolizumab, reslizumab, omalizumab, tezepelumab, or tralokinumab.
* Treatment with pramipexole (Mirapex®) within 30 days of the Baseline Visit.
* Treatment with selected drugs known to have a substantial risk of neutropenia in the past 30 days prior to the Screening Visit.
* Treatment with selected drugs known to have a substantial risk of QT prolongation in the past 30 days prior to the Screening Visit.
* Participants who are participating in the acute phase of a pulmonary rehabilitation program, ie, who started rehabilitation.
* History of malignancy that required surgery (excluding local and wide-local excision), radiation therapy and/or systemic therapy during the 2 years prior to the Baseline Visit.
* History of human immunodeficiency virus infection or chronic infection with hepatitis B or C.
* Neutrophil count <2.000x109/L at the Screening Visit.
* Renal dysfunction, defined as an estimated glomerular filtration rate <60 mL/min/1.73m2 at the Screening Visit (using the Chronic Kidney Disease Epidemiology Collaboration) formula.
* Active liver disease defined as any known current infectious, neoplastic, or metabolic pathology of the liver or unexplained elevations in alanine aminotransferase (ALT), aspartate aminotransferase (AST), >3x the upper limit of normal (ULN), or total bilirubin >2x ULN at the Screening Visit confirmed by a repeat abnormal measurement of the relevant value(s), at least 1 week apart.
* History of New York Heart Association class IV heart failure or last known left ventricular ejection fraction <25%.
* Corrected QT interval by Fridericia (QTcF) interval >450 ms for males and >470 ms for females at the Screening Visit or QTcF ≥480 ms for participants with bundle branch block.
* Pregnant women or women breastfeeding.
* Males who are unwilling to use an acceptable method of birth control during the entire study period (ie, condom with spermicide).
* The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-09 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Geometric mean change in the blood AEC from baseline to Week 16 | Baseline, Week 16

SECONDARY OUTCOMES:
Pre-BD FEV1 | Baseline, Week 16
  Change in pre-bronchodilator forced expiratory volume in 1 second (pre-BD FEV1) from baseline to Week 16
Post-BD FEV1 | Baseline, Week 16
  Change in post-bronchodilator forced expiratory volume in 1 second (Pre-BD FEV1) from baseline to Week 16
St George's Respiratory Questionnaire for COPD Patients (SGRQ-C) | Baseline, Week 16
  Change from baseline to Week 16. SGRQ-C total scores range from 0 to 100, with higher scores indicating more limitations.
COPD Assessment Test (CAT) | Baseline, Week 16
  Change from baseline to Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Gerard J Criner, MD, Principal Investigator — Temple University
Locations (23):
- United States (23):
  - Research Site US-10001-017, Conway, Arkansas
  - Research Site US-10001-008, Newport Beach, California
  - Research Site US-10001-022, Northridge, California
  - Research Site US-10001-016, Westminster, California
  - Research Site US-10001-030, Orlando, Florida
  - Research Site 10001-032, Champaign, Illinois
  - Research Site US-10001-021, Hammond, Indiana
  - Research Site US-10001-033, Des Moines, Iowa
  - Research Site US-10001-020, Baltimore, Maryland
  - Research Site US-10001-024, Farmington Hills, Michigan
  - Research Site US-10001-005, Saint Charles, Missouri
  - Research Site US-10001-001, St Louis, Missouri
  - Research US-10001-010, Charlotte, North Carolina
  - Research Site US-10001-025, Charlotte, North Carolina
  - Research Site US-10001-007, Gastonia, North Carolina
  - Research Site US-10001-004, Columbus, Ohio
  - Research Site US-10001-002, DuBois, Pennsylvania
  - Research Site US-10001-013, Philadelphia, Pennsylvania
  - Research Site US-10001-023, East Providence, Rhode Island
  - Research Site US-10001-012, Rock Hill, South Carolina
  - Research Site US-10001-009, Corsicana, Texas
  - Research Site US-10001-038, Houston, Texas
  - Research Site 10001-026, McKinney, Texas

IPD SHARING:
Plan to Share IPD: No